CLINICAL TRIAL: NCT05426460
Title: AAT + tDCS to Reduce Cue-induced Craving and Smoking Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynthia Conklin (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Cynthia Conklin, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY21020160; 1R21DA053395-01 (NIH)
Record Dates: First submitted 2022-05-26; First posted 2022-06-22 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-04

CONDITIONS: Smoking Behaviors; Smoking, Cigarette
Keywords: Transcranial Direct Current Stimulation (tDCS); Approach Avoidance Task (AAT); Smoking
MeSH Terms: conditions — Smoking; Cigarette Smoking | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The transcranial tDCS is delivered without the participant or investigator knowing if they are receiving tDCS or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- AAT + tDCS (Experimental): Approach Avoidance Task + Transcranial Direct Current Stimulation targeting the dorsolateral prefrontal cortex
  Interventions: Behavioral: Approach/Avoidance Task; Device: Transcranial Direct Current Stimulation
- AAT + sham tDCS (Sham Comparator): Approach Avoidance Task with Sham Transcranial Direct Current Stimulation.
  Interventions: Behavioral: Approach/Avoidance Task; Device: Sham tDCS
- AC + tDCS (Active Comparator): Active Control Task with Transcranial Direct Current Stimulation targeting the dorsolateral prefrontal cortex
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: AC
- AC + sham tDCS (Sham Comparator): Active Control Task with sham Transcranial Direct Current Stimulation
  Interventions: Behavioral: AC; Device: Sham tDCS

INTERVENTIONS:
Behavioral: Approach/Avoidance Task — The Approach/avoidance task (AAT) training is done using a joystick. The AAT tasks involves having participants push away pictures of smoking stimuli that appear on the screen by pushing the joystick forward, and pulling in pictures of nonsmoking stimuli that appear on the screen by pulling the joystick towards themselves. Pushing smoking-related pictures away causes the picture to shrink in size, whereas pulling a picture closer causes the picture to increase in size. This task consists of 4 blocks of 24 pictures, taking 30 minutes.
  Other Names: AAT
  Arms: AAT + sham tDCS; AAT + tDCS
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation active (2.0 mA) (tDCS) will be used to temporarily increase cortical excitability of the dorsolateral prefrontal cortex (dlPFC) in healthy daily smokers. Participants assigned to active tDCS conditions will receive active (2.0 mA) tDCS, with anode electrode placement over the right dlPFC and cathode electrode placement over the left bicep. tDCS will be administered the first 20 minutes of each of the five 30 minute AAT training sessions.
  Other Names: tDCS
  Arms: AAT + tDCS; AC + tDCS
Behavioral: AC — During Active Control (AC) participants press a button on the left of right of the joystick to indicate the position the picture on a screen. Position of pictures will be balanced across the 4 blocks of 24 pictures, taking 30 minutes.
  Arms: AC + sham tDCS; AC + tDCS
Device: Sham tDCS — Sham transcranial Direct Current Stimulation (0.1 mA) (sham tDCS) will be used as a control for active tDCS with anode electrode placement over the right dlPFC and cathode electrode placement over the left bicep. Sham tDCS will be administered during the first 20 minutes of each of the four blocks of 24 pictures, taking 30 minutes, across the 5 training sessions.
  Arms: AAT + sham tDCS; AC + sham tDCS

SUMMARY:
Smokers are highly reactive to smoking-related stimuli and report that this cue reactivity (CR) is a major obstacle to quitting. To date, no pharmacologic methods attenuate CR, and attempts to diminish it with traditional cue exposure treatment (CET) have not proven effective. The proposed study will test a highly novel cue-based smoking treatment adjunct combining an Approach/Avoidance Task (AAT) with brain stimulation via tDCS applied to the dorsolateral prefrontal cortex (dlPFC) during personalized multi-cue exposure; the goal of which is to discover an effective means of reducing cue reactivity and daily smoking, and increasing intent and confidence to quit, among high treatment-interest smokers.

DETAILED DESCRIPTION:
Exposure to smoking-related cues robustly increases self-report craving and immediate subsequent smoking. This cue-reactivity (CR) is an often-reported obstacle to quitting among smokers. Unlike methods to diminish abstinence-induced craving, which have been highly successful with the advent of nicotine replacement therapies (NRTs), pharmacotherapies have not been shown to diminish smoking-related reactivity to cues. Past behavioral methods to reduce smokers' CR, most commonly extinction training through cue-exposure treatment (CET), have also consistently failed. Review of past CET studies reveals that this failure is largely due to several methodological shortcomings including: (1) presenting only proximal cues (e.g., cigarettes, ashtrays), (2) conducting passive unreinforced exposure to these limited cues, and (3) achieving only limited new learning. The researchers extensive past cue work makes them uniquely qualified to remedy these flaws by designing and testing novel CET methodology incorporating contemporary techniques and technology to reduce CR and relieve smokers of this ubiquitous source of relapse risk. The researchers propose three methods to improve CET. First, using well-tested methods for personalizing smoking cues and presenting numerous proximal, environment, and people cues in combination, the proposed cue exposure will better capture and target the cue-rich situations most likely to trigger smokers' strongest CR. Second, rather than repeated passive unreinforced exposure to cues, smokers will engage in active re-training of approach biases toward their personal smoking stimuli using an Approach/Avoidance Task (AAT), a method shown to activate the dorsolateral prefrontal cortex (dlPFC), a brain region associated with both cognitive control over craving and deactivation of drug reward systems. Third, to enhance new learning, smokers will undergo non-invasive transcranial direct current brain stimulation (i.e., tDCS) of the dlPFC. Although the researchers propose each method, AAT and tDCS, should independently reduce smokers' CR to their most salient cues, providing AAT with simultaneous tDCS (AAT+tDCS) should synergistically attenuate CR by better increasing cortical excitability in the dlPFC. To assess this, a 2 x 2 active and sham-controlled test of AAT and tDCS during personalized multi-cue exposures will be used to examine pre-post training changes across several measures of smoking-related cue reactivity (cue-induced craving, cue-provoked smoking topography, and attentional bias measures of Evoked Response Potentials (ERPs) and reaction time), as well as changes in daily smoking and confidence and intent to quit pre-post training and at 1 week and 1-month follow up. The goal of this work is to develop an efficacious treatment adjunct that better prepares smokers to confront cues when they try to remain quit.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 26 & 55
* High treatment interest (planning to quit within the next 6 months)
* Ability to provide written informed consent
* Smoke equal or greater than 7 cigarettes per day
* Expired breath carbon monoxide (CO) equal or greater than 8 ppm at screening
* Ability to attend 10 sessions over a 3-week period, and complete 2 follow-up phone assessments

Exclusion Criteria:

* Epilepsy or Current Seizure Disorder
* Alcohol or Substance Dependence past 3 months (caffeine allowed, nicotine is part of inclusion criteria, alcohol > 14 drinks per week (M) or > 7 drinks per week (F))
* Implanted cardiac or brain medical devices
* History of epilepsy or current seizure disorder
* History of brain surgery or skull fracture
* History of a head trauma (losing consciousness >10 min and/or problems with speech or movement because of head injury)
* Latex allergy
* Scalp irritation
* History of diabetes that caused loss of consciousness (>10 min) or weakness in your arms or legs
* History of electroconvulsive therapy (ECT) in the last 5 years (Y / N) History of ECT within the last 5 years
* Current use of dextromethorphan
* Diagnosed with or undergone treatment for alcohol or substance dependence past 3 months
* Uncorrected vision deficit
* Colorblindness
* Use of tobacco products other than commercially available cigarettes

Ages: 26 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Conklin, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification may be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following publication, no end date
Access Criteria: Any purpose

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 04/29/2022 - 5/21/2024, 179 participants were screened via telephone call. 79 passed inital phone screening and attended an in-person session in the research laboratory in a medical hospital setting where a full inclusion criteria assessment was conducted.
Pre-assignment Details: Of the 79 participants who attended an inital in-person session for further screening, 23 chose not to participate in the study and 15 were deemed ineligble to continue. Forty-one participants signed informed consent and were randomized. However, 3 participants were excluded from the study after randomization leaving 38 participants contributing data and completing the study.
Period: Overall Study
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Started | 12 | 10 | 11 | 8
Completed | 11 | 9 | 10 | 8
Not Completed | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS | Total
Number analyzed (Participants) | 11 | 9 | 10 | 8 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 10 | 8 | 38
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (6.3) | 42.6 (8.7) | 45.8 (7.2) | 45.8 (7.9) | 44.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 5 | 4 | 19
  Male | 5 | 5 | 5 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 9 | 10 | 7 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 2 | 7
  White | 7 | 9 | 7 | 4 | 27
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 10 | 8 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in 4-item Questionnaire on Smoking Urges Craving Score During Cue Reactivity to Personal Cues
Description: Difference between cue-induced craving rating from pre-treatment (Baseline) to post-treatment (re-test) on the questionnaire on smoking urges 4-items scored 0-100. Lower values indicate more reduction in cue-induced craving.
Time Frame: Baseline to approximately 1 week
Population: 3 participants (2 from AAT + tDCS and 1 from AAT + sham tDCS) were excluded from analyses due to data collection error in which their ratings were not recorded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 9 | 8 | 10 | 8
score on a scale | -36.5 (20.0) | -36.3 (26.1) | -36.6 (34.2) | -22.2 (22.8)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 x 2 ANOVA; Test type: Superiority; p = .438, ANOVA

2. Primary Outcome: Mean Change From Baseline in Number Cigarettes Smoked Daily
Description: Difference in mean number of cigarette smoker per day from pre-treatment (Baseline) to post-treatment (re-test). Lower number indicates greater reduction in cigarettes smoked.
Time Frame: Baseline to approximately 1 week
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 11 | 10 | 9 | 8
cigarettes per day | -3.6 (3.1) | -2.6 (4.7) | -2.1 (5.9) | -0.4 (6.5)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 x 2 ANOVA; Test type: Superiority; p = .847, ANOVA

3. Primary Outcome: Mean Change From Baseline in Number Cigarettes Smoked Daily
Description: Difference in mean number of cigarettes smoked per day from pre-treatment (Baseline) to 1 week post treatment (follow-up). Lower number indicates greater reduction in cigarettes smoked.
Time Frame: Baseline to approximately 2 weeks
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 11 | 9 | 10 | 8
cigarettes per day | -3.9 (2.4) | -3.3 (5.7) | -1.7 (5.4) | -3.0 (6.9)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 X 2 ANOVA; Test type: Superiority; p = .570, ANOVA

4. Primary Outcome: Mean Change From Baseline in Number Cigarettes Smoked Daily
Description: Difference in mean number of cigarette smoker per day from pre-treatment (Baseline) to 1 month post treatment (follow-up). Lower number indicates greater reduction in cigarettes smoked.
Time Frame: Baseline to approximately 6-weeks
Population: 3 participants (1 from AAT + tDCS, 1 from AA + sham tDCS, and 1 from AC + tDCS) were lost to follow-up.
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 10 | 8 | 9 | 8
cigarettes per day | -3.8 (3.9) | -5.5 (3.8) | -4.3 (5.9) | -4.6 (5.0)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 x 2 ANOVA; Test type: Superiority; p = .657, ANOVA

5. Primary Outcome: Mean Change From Baseline in Rating Score for 5-item Confidence to Quit Questionnaire
Description: Difference between Confidence to Quit score from pre-treatment (Baseline) to post-treatment (re-test) scored 0-100. More positive score reflects an increase in confidence to quit smoking.
Time Frame: Baseline to approximately 1-week
Population: Data is missing from 2 participants (1 from AAT + tDCS and 1 from AC + sham tDCS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 10 | 9 | 10 | 7
score on a scale | 1.0 (18.0) | 8.9 (20.0) | 3.0 (18.6) | 27.1 (24.3)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 x 2 ANOVA; Test type: Superiority; p = .254, ANOVA

6. Primary Outcome: Mean Change From Baseline in Rating Score for 5-item Confidence to Quit Questionnaire
Description: Difference between Confidence to Quit rating from pre-treatment (Baseline) to 1 week post-treatment (follow-up)
Time Frame: Baseline to approximately 2-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 11 | 9 | 10 | 8
score on a scale | -4.4 (28.4) | 6.9 (20.4) | 6.6 (17.8) | 20.0 (23.1)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 x 2 ANOVA with Main effect p-values for tDCS and AAT reported in comments below; Test type: Superiority; p = .852, ANOVA

7. Primary Outcome: Mean Change From Baseline in Rating Score for 5-item Confidence to Quit Questionnaire
Description: Difference between Confidence to Quit rating from pre-treatment (Baseline) to 1 month post-treatment (follow-up)
Time Frame: Baseline to approximately 6-weeks
Population: 3 participants were lost to follow up (1 each in groups AAT + tDCS, AAT + sham tDCS, and AC+tDCS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 10 | 8 | 9 | 8
score on a scale | 2.8 (24.5) | 13.3 (20.0) | 12.2 (22.4) | 22.8 (24.8)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 x 2 ANOVA; Test type: Superiority; p = .732, ANOVA

8. Primary Outcome: Mean Change From Baseline in Rating Score for Intent to Quit Questionnaire
Description: Difference between Intent to Quit score from pre-treatment (Baseline) to post-treatment (re-test). Scale is rated 1-10 from 1= "I have no thoughts about or interest in quitting smoking" to 10= "I have quit and will never go back" A positive change score indicates an increased intention to quit.
Time Frame: Baseline to approximately 1-week
Population: 2 participants are not included in the analyses due to missing data (1 from AAT + tDCS, 1 from AC + sham tDCS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 10 | 9 | 10 | 7
score on a scale | 1.2 (1.0) | 0.4 (0.9) | -0.2 (0.8) | 0.7 (1.6)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 x 2 ANOVA; Test type: Superiority; p = .038, ANOVA

9. Primary Outcome: Mean Change From Baseline in Rating Score for Intent to Quit Questionnaire
Description: Difference between Intent to Quit score from pre-treatment (Baseline) to 1 week post-treatment (follow-up). Scale is rated 1-10 from 1= "I have no thoughts about or interest in quitting smoking" to 10= "I have quit and will never go back" A positive change score indicates an increased intention to quit.
Time Frame: Baseline to approximately 2-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 11 | 9 | 10 | 8
score on a scale | 1.3 (1.2) | 0.9 (0.6) | -0.3 (0.9) | 1.1 (1.5)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 x 2 ANOVA; Test type: Superiority; p = .029, ANOVA

10. Primary Outcome: Mean Change From Baseline in Rating Score for Intent to Quit Questionnaire
Description: Difference between Intent to Quit score from pre-treatment (Baseline) to 1 month post-treatment (follow-up). Scale is rated 1-10 from 1= "I have no thoughts about or interest in quitting smoking" to 10= "I have quit and will never go back" A positive change score indicates an increased intention to quit.
Time Frame: Baseline to approximately 6-weeks
Population: Data from 3 participants (1 from AAT + tDCS, 1 From AAT + sham tDCS, and 1 from AC + tDCS) were lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
Number analyzed (Participants) | 10 | 8 | 9 | 8
score on a scale | 1.4 (1.3) | 1.3 (1.4) | 0.6 (1.7) | 1.3 (1.8)
Statistical Analysis 1: Comparison: AAT + tDCS vs AAT + Sham tDCS vs AC + tDCS vs AC + Sham tDCS; 2 x 2 ANOVA; Test type: Superiority; p = .353, ANOVA

ADVERSE EVENTS:
Time Frame: Tracking of adverse occurred over 2 years, 1 month
Arm/Group | AAT + tDCS | AAT + Sham tDCS | AC + tDCS | AC + Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/11 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT05426460/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT05426460/ICF_000.pdf